CLINICAL TRIAL: NCT01114555
Title: Combination of Bevacizumab, Irinotecan and Temozolomide for Relapsed or Refractory Neuroblastoma: A Phase II Study
Brief Title: Bevacizumab, Irinotecan and Temozolomide for Relapsed or Refractory Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-015
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2018-11

CONDITIONS: Neuroblastoma
Keywords: Bevacizumab; Irinotecan; Temozolomide; 10-015
MeSH Terms: conditions — Neuroblastoma | interventions — Bevacizumab; Irinotecan; Temozolomide

ARMS (1):
- Bevacizumab, Irinotecan and Temozolomide (Experimental): This is a phase II study of the combination of irinotecan, temozolomide and bevacizumab in patients with resistant NB.
  Interventions: Drug: Bevacizumab, Irinotecan and Temozolomide

INTERVENTIONS:
Drug: Bevacizumab, Irinotecan and Temozolomide — Patients will initially receive bevacizumab IV at 15mg/kg/dose (this is defined as Day 1 Three days later (starting day 4), they will receive concurrently, IV irinotecan at 50mg/m2/day x 5 days plus PO temozolomide 150mg/m2/day x 5 days. A second dose of bevacizumab will be administered 14 days after the first one(day 15). The treatment schedule may require minor adjustment as clinically indicated (e.g., due to PDH closure for holidays).

SUMMARY:
The purpose of this study is to find how good and how safe the combination of irinotecan, temozolomide and bevacizumab is for patients with resistant or recurrent neuroblastoma. These drugs have each been given separately to patients, but they have never been given all together. Irinotecan and temozolomide are two drugs that have been used together to treat neuroblastoma in many people. These drugs are considered chemotherapy. Bevacizumab is another drug used to treat cancer. It is made by a company called Genentech. Bevacizumab is an antibody. Antibodies are proteins that are found in the blood and can attach themselves to bacteria and viruses. Bevacizumab attaches itself to a special protein in the bloodstream. This protein helps tumors grow new blood vessels. Blood vessels carry nutrients to feed the tumor. Bevacizumab is thought to block this growth of new blood vessels and starve tumors. It has been used for the treatment of many cancers in adults. It is approved by the FDA for the treatment of adults with colon cancer and other cancers but not for people with neuroblastoma. There is only a small amount of information known on using this drug in children. It has been used with irinotecan before to treat cancer but not in children with neuroblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the diagnosis of NB in accordance with the International Criteria, i.e., either histopathology (confirmed by the MSKCC Department of Pathology) or BM involvement plus elevated urinary catecholamines.
* Must have a history of tumor progression or recurrence or failure to achieve complete response with standard therapy.
* Patients must have evaluable (microscopic marrow metastasis, MIBG or PET scans) or measurable (CT, MRI) disease.
* Patients of all ages are eligible.
* Prior Therapy: At least 2 weeks should have elapsed since any biologic therapy. Three weeks should have elapsed since last dose of chemotherapy.
* Minimum life expectancy of eight weeks.
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Severe major organ toxicity. Renal, cardiac, hepatic, pulmonary, gastrointestinal and neurologic toxicity should all be grade 2 or less (per NCI CTC version 4.0 criteria). Specifically, serum creatinine should be ≤3 x upper limit of normal (ULN), serum AST and ALT ≤5 x ULN, serum bilirubin ≤ 3 x ULN, LV shortening fraction should be ≥15%.
* Patients with myelosuppression are not excluded if ANC ≥ 500/uL. Platelet count should be > 35,000/ul and hemoglobin should be > 8gm/dl. Patients should not have received filgrastim, platelet or red blood cell transfusions for 2 days prior to achieving the above ANC, platelet and hemoglobin levels.
* Patients with documented chronic non-healing wound, ulcer or bone fracture
* Surgical procedures.
* Patients who have undergone major surgery <28 days prior to beginning therapy with bevacizumab are excluded.
* Patients must be least 24 hours from having after surgical procedures such as placement of central catheter.
* Patients <7days from minor surgeries (e.g. fine needle or core biopsies) and/or the unhealed wounds from these procedures are excluded.
* Patients will be excluded if major surgery (e.g. abdominal or thoracic surgery for resection of tumor) is anticipated during the course of the study.
* Known bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* Thrombosis: patients must not have had a deep venous or arterial thrombosis (non-central venous catheter related) within the last three months prior to study entry. Patients with cerebrovascular accident or transient ischemic attack within 6 months of therapy are excluded. Patients with history of peripheral vascular disease, myocardial infarction or unstable angina are excluded.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study entry.
* Known CNS metastases, except for treated brain metastasis. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement except for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include radiotherapy, chemotherapy or immunotherapy Patients with CNS metastases treated by neurosurgical resection or biopsy performed within 3 months of treatment will be excluded.
* Proteinuria: Urine protein: creatinine ratio ≥ 1.0.
* Uncontrolled (lasting >24 hrs on antihypertensive medication) hypertension as defined by age-appropriate criteria. Hypertension is defined as average systolic blood pressure and/or diastolic blood pressure that is 95th percentile for gender, age, and height on 3 occasions93. 95th percentiles for gender, age and height are provided in Appendix A. For patients ≥18 years of age, hypertension is defined as systolic blood pressure >150mmHg and/or diastolic blood pressure >100mmHg.
* Prior history of hypertensive crisis or hypertensive encephalopathy
* History of hypersensitivity to any component of bevacizumab
* History of hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1.
* Active serious infections not controlled by antibiotics.
* Pregnant women are excluded for fear of danger to the fetus. Therefore negative pregnancy test is required for all women of child-bearing age, and appropriate contraception is used during the study period.
* Inability or unwillingness to comply with protocol requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-04-29 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shakeel Modak, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Modak S, Kushner BH, Basu E, Roberts SS, Cheung NK. Combination of bevacizumab, irinotecan, and temozolomide for refractory or relapsed neuroblastoma: Results of a phase II study. Pediatr Blood Cancer. 2017 Aug;64(8):10.1002/pbc.26448. doi: 10.1002/pbc.26448. Epub 2017 Jan 23. PMID 28111925
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab, Irinotecan and Temozolomide
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab, Irinotecan and Temozolomide
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 6 [1 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Responses
Description: To evaluate tumor responses to combination of irinotecan, temozolomide and bevacizumab in patients with resistant NB.
Time Frame: 15-35 days after cycle 2
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab, Irinotecan and Temozolomide
Number analyzed (Participants) | 34
Participants
  Complete Response | 3
  No Response | 18
  Progressive Disease | 12
  Not Treated | 1

2. Secondary Outcome: Number of Participants With Treatment Related Toxicity
Description: To determine the toxicity of the combination of irinotecan, temozolomide and bevacizumab in patients with resistant NB.
Time Frame: Patients will be evaluated at least once weekly for toxicity. Observation for toxicities for up to 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab, Irinotecan and Temozolomide
Number analyzed (Participants) | 34
Participants | 34

3. Secondary Outcome: To Evaluate Changes in Angiogenic Markers After Treatment With the Combination of Irinotecan, Temozolomide and Bevacizumab.
Time Frame: days 1,4, 15 and once between days 22-35 during cycle 1 and cycle 2
Population: Data were not collected
Arm/Group | Bevacizumab, Irinotecan and Temozolomide
Number analyzed (Participants) | 0

4. Secondary Outcome: To Measure Time to Progression in Patients With Resistant NB Treated With the Combination of Irinotecan, Temozolomide and Bevacizumab.
Time Frame: 3 years
Population: Data were not collected
Arm/Group | Bevacizumab, Irinotecan and Temozolomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Bevacizumab, Irinotecan and Temozolomide
All-Cause Mortality (participants affected / at risk) | 27/34
Serious Adverse Events (participants affected / at risk) | 14/34
Other Adverse Events (participants affected / at risk) | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab, Irinotecan and Temozolomide (N=34)
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 2
Chills (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Enterocolitis infectious (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Seizure (Nervous system disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab, Irinotecan and Temozolomide (N=34)
Thrombocytopenia (Investigations) | 31
Neutropenia (Blood and lymphatic system disorders) | 29
Lymphopenia (Investigations) | 28
Diarrhea (Gastrointestinal disorders) | 27
Elevated AST (Investigations) | 26
Elevated ALT (Investigations) | 21
Vomiting (Gastrointestinal disorders) | 19
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 4
Proteinuria (Renal and urinary disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT01114555/Prot_SAP_000.pdf